CLINICAL TRIAL: NCT02304393
Title: An Open-Label, Multicenter, Dose-Escalation Phase IB Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Therapeutic Activity of Selicrelumab (CD40 Agonist) in Combination With Atezolizumab (Anti PD-L1) in Patients With Locally Advanced and/or Metastatic Solid Tumors
Brief Title: A Study of Selicrelumab (RO7009789) in Combination With Atezolizumab in Participants With Locally Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP29392; 2014-002835-32 (EudraCT Number)
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab; selicrelumab

ARMS (4):
- Part IA: Selicrelumab (IV) + Atezolizumab (Experimental): Selicrelumab at a dose of 16 milligrams (mg) will be administered intravenously (IV) on Day 1 of Cycle 1 (first cycle in this group was of 42 days, and subsequent 21-day cycles); and atezolizumab 1200 mg will be administered IV after 6 weeks on Day 1 of Cycle 2, followed by every 3 weeks during Part IA until disease progression, death, loss of follow-up, or withdrawal of consent.
  Interventions: Drug: Atezolizumab; Drug: Selicrelumab
- Part IA: Selicrelumab(SC) + Atezolizumab (Experimental): Selicrelumab at a starting dose of 1 mg will be administered subcutaneously (SC) on Day 1 of Cycle 1 (21-day cycle) which will follow escalation in sequential cohorts; and atezolizumab 1200 mg will be administered IV on Day 1 of Cycle 2, and followed by every 3 weeks during Part IA as long as the participant experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Selicrelumab
- Part IB: Selicrelumab + Atezolizumab (Experimental): Selicrelumab will be administered at a starting dose of 1 mg SC on Day 2 of Cycle 1 (21-day cycle) which will follow escalation in sequential cohorts; and atezolizumab 1200 mg will be administered IV on Day 1 of Cycle 1, and followed by every 3 weeks during Part IB as long as the participant experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Selicrelumab
- Part II: Selicrelumab + Atezolizumab (Experimental): Atezolizumab 1200 mg will be administered IV on Day 1 of Cycle 1, and followed by every 3 weeks; and Selicrelumab will be administered at the dose defined in Part IB (not exceeding 80 mg SC [unless IV administration in Part IB demonstrates better benefit/risk ratio]) on Day 2 (1 day after atezolizumab administration) of every second cycle from Cycles 1 to 7, and every fourth cycle thereafter during Part II as long as the participant experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Selicrelumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as per the dosage regimen mentioned in respective arm descriptions.
  Other Names: MPDL3280A; Tecentriq
Drug: Selicrelumab — Selicrelumab will be administered as per the dosage regimen mentioned in respective arm descriptions.
  Other Names: RO7009789

SUMMARY:
This is an open-label, multicenter study designed to assess the safety, pharmacokinetics, pharmacodynamics and activity of Selicrelumab administered in combination with Atezolizumab (ATZ) in participants with metastatic or locally advanced solid tumors. The study will be conducted in two Parts (I and II), with Part I divided into Parts IA and IB. All participants will be followed up for survival until death or loss of follow-up after the last visit or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of locally advanced and/or metastatic solid tumors, which are not amenable to standard therapy
* Part I: histologically confirmed diagnosis of advanced/metastatic small and large bowel carcinomas (small bowel and CRC), CPI-experienced non-small cell lung cancer (NSCLC) and head and neck squamous cell carcinoma (HNSCC)
* Part II: CPI-experienced NSCLC patients must have experienced documented disease progression on or after PD-L1 or PD-1 inhibitor therapy (investigational or approved): screening tumor assessment should confirm prior progression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 16 weeks
* Adequate hematologic and end organ function
* Measurable disease per RECIST Version 1.1
* Ability to comply with the protocol requirements
* Female participants of childbearing potential must have a negative pregnancy test (urine/serum) within seven days prior to the first study drug administration
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1% per year during the treatment period and for at least 5 months after the last dose of study treatment
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for at least 28 days after the last dose of study treatment

Exclusion Criteria:

* If one of the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1 Day 1) are: soluble interleukin 2 receptor (sCD25) greater than (>) 2 × upper limit of normal (ULN); Serum ferritin >1000 nanograms per milliliter (ng/mL)
* Any approved anti-cancer therapy that includes chemotherapy, hormonal therapy, or radiotherapy within 2 weeks prior to the first dose of study treatment; the following is, however, allowed: Palliative radiotherapy for bone metastases less than or equal to (</=) 2 weeks prior to Cycle 1 Day 1
* Adverse events from prior anti-cancer therapy that have not resolved to Grade </= 1 except for any grade alopecia and </= Grade 2 peripheral neuropathy
* Bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (example: bone metastasis or osteoporosis) is allowed
* Uncontrolled pleural effusion, pericardial effusion, or ascites that require recurrent drainage procedures (one monthly or more frequently). Participants with indwelling catheters are allowed
* Known clinically significant liver disease which includes active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
* History (within the previous year) of congestive heart failure, stroke, arrhythmia, or myocardial infarction
* History of peripheral venous thrombosis or thromboembolic event (within 12 months prior to Cycle 1 Day 1)
* Significant cardio- or cerebrovascular disease within 6 months prior to Cycle 1 Day 1
* Known hereditary or acquired coagulopathies
* Clinically meaningful proteinuria
* Requiring dialysis (peritoneal or hemodialysis)
* Known primary central nervous system (CNS) malignancy or symptomatic or untreated CNS metastases: participants with asymptomatic-treated CNS metastases may be enrolled after consultation with the Medical Monitor, provided they meet the following criteria:

  1. Radiographic demonstration of improvement upon completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
  2. No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1 Day 1
* Pregnancy, lactation, or breastfeeding
* Allergy or hypersensitivity to components of the RO7009789 formulation or to components of atezolizumab formulation
* History of autoimmune diseases (participants with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible; participants with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study)
* History of idiopathic pulmonary fibrosis, pneumonitis (excluding infectious disease-induced), organizing pneumonia, or evidence of active pneumonitis
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Participants with human immunodeficiency virus (HIV) infection, active hepatitis B (chronic or acute), or hepatitis C infection
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1 Day 1
* Signs or symptoms of infection within 2 weeks prior to Cycle 1 Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* Major surgical procedure within 28 days prior to Cycle 1 Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Malignancies other than disease under study within 3 years prior to Cycle 1 Day 1 with the exception of those with a negligible risk of metastasis or death and with expected curative outcome
* Previous treatment with any other compound that targets cluster of differentiation 40 (CD40) (like Chi Lob 7/4 and ADC1013)
* Treatment with systemic immunostimulatory agents (including but not limited to interferon (IFN)-alpha, Interleukin-2 (IL-2) within 4 weeks or 5 times the half-life of the drug, whichever is shorter, prior to Cycle 1 Day 1
* Treatment with investigational agent within 4 weeks prior to Cycle 1 Day 1 (or within 5 times the half-life of the investigational product, whichever is longer)
* Concomitant treatment with anticoagulants (example: coumadin, heparin) except low dose molecular weight heparin for prophylactic purposes and direct factor Xa inhibitors
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF) agent within 2 weeks prior to Cycle 1 Day 1

  1. Participants who have received acute, low-dose, systemic immunosuppressant medications (example: a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Medical Monitor
  2. The use of corticosteroids as premedication in case of dye allergy previous to computed tomography (CT) scan is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participants at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Part IA: Percentage of Participants with Adverse Events and Serious Adverse Events | Baseline up to 28 Days After the Last Dose (Approximately 38 Months)
Part IB: Percentage of Participants with Adverse Events and Serious Adverse Events | Baseline up to 28 Days After the Last Dose (Approximately 38 Months)
Part IB: Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Cycle 1 Day 1 up to Cycle 2 Day 2 (Cycle length = 21 days)
Part IB: Maximum Tolerated Dose (MTD) of Selicrelumab | Cycle 1 Day 1 up to Cycle 2 Day 2 (Cycle length = 21 days)
Part IB: Recommended Part II Dose of Selicrelumab | Cycle 1 Day 1 up to Cycle 2 Day 2 (Cycle length = 21 days)
Part II: Percentage of Participants with Adverse Events and Serious Adverse Events | Baseline up to 28 days after the last dose (approximately 38 months)
Part II: Percentage of Participants With Best Overall Response, as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Progression-Free Survival (PFS), as Determined by Investigator Using RECIST Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Duration of Objective Response, as Determined by Investigator Using RECIST Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Percentage of Participants With Disease Control, as Determined by Investigator Using RECIST Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Percentage of Participants With Disease Control, as Determined by Investigator Using Unidimensional irRC | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: PFS, as Determined by Investigator Using Unidimensional irRC | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Percentage of Participants With Best Overall Response, as Determined by Investigator Using Unidimensional Immune-Related Response Criteria (irRC) | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Duration of Objective Response, as Determined by Investigator Using Unidimensional irRC | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Overall Survival | Baseline up to death due to any cause (up to approximately 38 months)

SECONDARY OUTCOMES:
Part IA: Area Under the Concentration Time Curve (AUC) of Selicrelumab | Pre Selicrelumab dose (1hour[Hr]) on Cycle(Cy)1 Day1(D1); 4,8,24,48,72Hr post D1dose; D8,15 of Cy1; D1 Cy2&3 (10 minutes pre ATZ dose); at radiographic disease progression (PD)(up to 38 months);28&150 days after last ATZ dose (up to38months)(Cy=21days)
Part IA: Maximum Serum Concentration (Cmax) of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 minutes [min] pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IA: Time to Cmax (Tmax) of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IA: Minimum Serum Concentration Under Steady-State (Cmin) of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IA: Apparent Clearance (CL/F) of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IA: Half-Life (t1/2) of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IA: Cmax of Atezolizumab | Pre ATZ (within 10 min) & at end of 60 min ATZ infusion on Cy2D1; pre ATZ dose (within 10 min) on D1 of Cy3,4,5,9,& every 8Cy thereafter(up to 38 months); at radiographic PD(up to 38 months); 28&150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IA: Cmin of Atezolizumab | Pre ATZ (within 10 min) & at end of 60 min ATZ infusion on Cy2D1; pre ATZ dose (within 10 min) on D1 of Cy3,4,5,9,& every 8Cy thereafter(up to 38 months); at radiographic PD(up to 38 months); 28&150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: AUC of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Cmax of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Tmax of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Cmin of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: CL/F of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Apparent Volume of Distribution (V/F) of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: t1/2 of SC Selicrelumab | Pre ATZ dose (within 1 Hr) on Cy1D1, Pre Selicrelumab dose (within 1 Hr) on Cy1D2; Cy1 D3,4,5,9,15 post D2 dose; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Cmax of Atezolizumab | Pre ATZ (within 1 Hr) & at end of 60 min ATZ infusion on Cy1D1; pre ATZ dose (within 10 min) on D1 of Cy2,3,4,8,& every 8Cy thereafter (up to 38 months); at radiographic PD (up to 38 months); 28&150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part IB: Cmin of Atezolizumab | Pre ATZ (within 1 Hr) & at end of 60 min ATZ infusion on Cy1D1; pre ATZ dose (within 10 min) on D1 of Cy2,3,4,8,& every 8Cy thereafter (up to 38 months); at radiographic PD (up to 38 months); 28&150 days after last ATZ dose (up to 38 months) (Cy=21 days)
Part II: AUC of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy1,5D5,8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2 of Cy3,5,11,15,19; D8 of Cy11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: Cmax of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy1, 5D5, 8, 15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2-Cy3,5,11,15,19; D8-Cy 11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: Tmax of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy 1, 5 D5,8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2 of Cy3,5,11,15,19; D8 of Cy 11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: Cmin of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy1,5D5, 8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy11, 15, 19; pre Selicrelumab(10 min) on D2-Cy3,5,11,15,19; D8-Cy 11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: CL/F of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy1,5D5,8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2-Cy3,5,11,15,19; D8-Cy11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: V/F of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy 1,5D5,8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2-Cy3,5,11,15,19; D8-Cy 11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: t1/2 of Selicrelumab | Pre Selicrelumab (within 1Hr) on Cy1D2; Cy1,5D5,8,15; pre ATZ (10 min) on D1-Cy2,4,6,8 and thereafter except Cy 11, 15, 19; pre Selicrelumab(10 min) on D2-Cy3,5,11,15,19; D8-Cy 11,15,19; 28&150 days after last ATZ (up to 38 months) (Cy=21days)
Part II: Cmax of Atezolizumab | Cy1D1: pre ATZ dose (within 1 Hr), at end of ATZ infusion (60 min infusion); pre-ATZ dose (within 10 min)on D1 Cy2, 3, 4, 5, 6, 8, and thereafter (up to 38 months); 28 and 150 days after last ATZ dose (up to 38 months) (Cy = 21 days)
Part II: Cmin of Atezolizumab | Cy1D1: pre ATZ dose (within 1 Hr), at end of ATZ infusion (60 min infusion); pre-ATZ dose (within 10 min)on D1 Cy2, 3, 4, 5, 6, 8, and thereafter (up to 38 months); 28 and 150 days after last ATZ dose (up to 38 months) (Cy = 21 days)
Part IB: Percentage of Participants With Best Overall Response, as Determined by Investigator Using Unidimensional Immune-Related Response Criteria (irRC) | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part IB: Percentage of Participants With Best Overall Response, as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part IB: Percentage of Participants With Disease Control, as Determined by Investigator Using RECIST Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part Ib: Percentage of Participants With Disease Control, as Determined by Investigator Using Unidimensional irRC | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part IB: Duration of Objective Response, as Determined by Investigator Using RECIST Version 1.1 | First occurrence of response up to relapse or death due to any cause, whichever occurs first (up to approximately 38 months)
Part Ib: Duration of Objective Response, as Determined by Investigator Using Unidimensional irRC | First occurrence of response up to relapse or death due to any cause, whichever occurs first (up to approximately 38 months)
Part IB: Progression-Free Survival (PFS), as Determined by Investigator Using RECIST Version 1.1 | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part IA, IB, and II: Percentage of Participants With Auto-antibodies | Pre Selicrelumab dose(within 1 Hr) on Cy1D1;pre ATZ dose(within 10 min) on D1 Cy2,3,4,5 and every 8 cycles thereafter, up to 38 months); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months overall) (Cy=21 days)
Part IA, IB, and II: Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to Selicrelumab | Pre Selicrelumab dose(within 1 Hr) on Cy1D1;pre ATZ dose(within 10 min) on D1 Cy2,3,4,5 and every 8 cycles thereafter, up to 38 months); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months overall) (Cy=21 days)
Part IA, IB, and II: Percentage of Participants With ATA to ATZ | Pre ATZ(within 10 min)on D1 Cy2,3,4,5(Part IA),9(Cy8 for Part II)& every 8 cycles thereafter(up to 38 months);pre ATZ(within 1Hr) on Cy1D1(for Part IB & II);at radiographic PD(up to 38 months),28&150 days after last ATZ dose(up to 38 months)(Cy=21 days)
Part IA: Levels of Circulating Ki67 T cells Assessed by Immunophenotyping by Flow Cytometry | Cy1 D1: predose Selicrelumab D4 D8 D15 Cy2 D1: predose Atezo D3 D8 Cy3 D1: predose Atezo D8 PD at IRR/ISR (Cy=21 Days)
Part IB: Levels of Circulating Ki67 T Cells Assessed by Immunophenotyping by Flow Cytometry | Cy1: D3 D4 D5 D9 D15; Cy2: D1 D8; Cy4-47: D1 PD at IRR/ISR (Cy = 21 days)
Part II: Levels of Circulating Ki67 T Cells Assessed by Immunophenotyping by Flow Cytometry | Cy1: D1 pre-Atezo, D8, D15; Cy2D1: pre-Atezo; Cy3 D1 pre-Atezo, D8; Cy4D1: pre-Atezo; Cy5: D1 pre-Atezo, D8, D15; Cy6D1: Pre-Atezo; Cy11, 15 and 19: D1 pre Atezo and D8; After last Atezo dose SFU at IRR/ISR (Cy= 21 Days)
Part IA: Levels of Cluster of Differentiation 8 (CD8+) Cells Tumor-Infiltration Assessed by Immunophenotyping by Flow Cytometry | Cy1 D1: predose Selicrelumab D4 D8 D15; Cy2 D1: predose Atezo D3 D8; Cy3 D1: predose Atezo D8 PD at IRR/ISR (Cy= 21 Days)
Part IB: Levels of CD8+ Cells Tumor-Infiltration Assessed by Immunophenotyping by Flow Cytometry | Cy1: D1 predose, D3, D4, D5, D9, D15; Cy2: D1 predose, D8; Cy4-47: D1 predose, PD at IRR/ISR (Cy = 21 days)
Part IA: Levels of Programmed Death Ligand 1 (PD-L1) Expression on Both Tumor and Immune-Infiltrating Cells Assessed by Immunophenotyping by Flow Cytometry | Cy1 D1: predose Selicrelumab D4 D8 D15; Cy2 D1: predose Atezo D3 D8; Cy3 D1: predose Atezo D8 PD at IRR/ISR (Cycle = 21 Days)
Part IB: Levels of PD-L1 Expression on Both Tumor and Immune-Infiltrating Cells Assessed by Immunophenotyping by Flow Cytometry | Cy1: D1 predose, D3, D4, D5, D9, D15; Cy2: D1 predose, D8; Cy4-47: D1 predose, PD at IRR/ISR (Cy = 21 days)
Part II: Levels of PD-L1 Expression on Both Tumor and Immune-Infiltrating Cells Assessed by Immunophenotyping by Flow Cytometry | Cy1: D1 pre-Atezo, D8, D15; Cy2D1: pre-Atezo; Cy3 D1 pre-Atezo, D8; Cy4D1: pre-Atezo; Cy5: D1 pre-Atezo, D8, D15; Cy6D1: Pre-Atezo; Cy11, 15 and 19: D1 pre-Atezo and D8; After last Atezo dose SFU at IRR/ISR (Cy= 21 Days)
Part IA: V/F of Selicrelumab | Pre Selicrelumab dose (within 1 Hr) on Cy1 D1; 4, 8, 24, 48,72Hr post D1dose; D8, D15 of Cy1; D1 of Cy2 & 3 (10 min pre ATZ dose); at radiographic PD (up to 38 months); 28 & 150 days after last ATZ dose (up to 38 months) (Cy=21days)
Part IB: PFS, as Determined by Investigator Using Unidimensional irRC | Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 38 months)
Part II: Levels of CD8+ Cells Tumor-Infiltration Assessed by Immunophenotyping by Flow Cytometry | Part II: Pre ATZ (within 1 Hr) Cy1, 6, 11, 15, 19 D1; Cy1 D8, 15; pre ATZ (within 10 min) Cy2, 3, 4, 5 D1; Cy3, 5, 11, 15, 19 D8; Cy 5 D15; 28 days after last ATZ dose(up to 38 months); at radiographic tumor regression/PD (up to 38 months) (Cy= 21 days)
Part IB: AUC of IV Selicrelumab | Pre ATZ(1 Hr) Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mon)(Cy=21days)
Part IB: Cmax of IV Selicrelumab | Pre ATZ(1 Hr)Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mont)(Cy=21days)
Part IB: Cmin of IV Selicrelumab | Pre ATZ(1 Hr) Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mon)(Cy=21days)
Part IB: Total Clearance (CL) of IV Selicrelumab | Pre ATZ(1 Hr) Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mon)(Cy=21days)
Part IB: Volume of Distribution (Vss) of IV Selicrelumab | Pre ATZ(1 Hr) Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mon)(Cy=21days)
Part IB: t1/2 of IV Selicrelumab | Pre ATZ(1 Hr) Cy1D1,2;end of 30-min Selicrelumab infusion,0.25,2,4,6,8,10Hr post infusion start Cy1D2;24,30-36,48,72Hr Post Cy1D2 dose;Cy 1D9;D1 Cy2,3(10min pre ATZ);at radiographic PD(up to 38mon);28&150days after last ATZ dose(up to38mon)(Cy=21days)
Part IA: Percentage of Participants with Incidence of ADA Responses to RO7009789 | Pre-Dose Day 1 on Cycles 1, 2, 3, 4, 7 (Cycle length = 21 days); Safety Follow-up Visit (Up to 52 Days Post Final Dose)
Part IA: Percentage of Participants with Incidence of ADA Responses to Vanucizumab | Pre-Dose Day 1 on Cycles 1, 2, 4, 6, 8 (Cycle length = 21 days); Safety Follow-up Visit (Up to 52 Days Post Final Dose)
Part IB: Percentage of Participants with Incidence of ADA Responses to RO7009789 | Pre-Dose Day 1 on Cycles 1, 2, 3, 4, 7 (Cycle length = 21 days); Safety Follow-up Visit (Up to 52 Days Post Final Dose)
Part IB: Percentage of Participants with Incidence of ADA Responses to Vanucizumab | Pre-Dose Day 1 on Cycles 1, 2, 4, 6, 8 (Cycle length = 21 days); Safety Follow-up Visit (Up to 52 days post final dose)
Part II: Percentage of Participants with Incidence of ADA Responses to RO7009789 | Pre-Dose Day 1 on Cycles 1, 2, 3, 4, 7 (Cycle length = 21 days); Safety Follow-up Visit (Up to 52 Days Post Final Dose)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Canada (2):
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Jewish General Hospital / McGill University, Montreal, Quebec
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- France (3):
  - Aphm; Cpcet, Marseille
  - Hopital Saint Louis, Service D Oncologie Medicale, Paris
  - Institut Gustave Roussy; Sitep, Villejuif
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Medisch Centrum Rotterdam; Lokatie Daniel den Hoed, Rotterdam
- Spain (2):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid